CLINICAL TRIAL: NCT07048249
Title: Single Arm Evaluation of Romiplostim to Prevent Chemotherapy Induced Thrombocytopenia in Patients With Ewing Sarcoma
Brief Title: Single Arm Romiplostim to Prevent CIT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Romiplostim-BT-2201
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Ewings Sarcoma; Chemotherapy Induced Thrombocytopenia
Keywords: romiplostim; ewing sarcoma; chemotherapy induced thrombocytopenia; CIT; NPLATE
MeSH Terms: conditions — Sarcoma, Ewing | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Romiplostim administration with chemotherapy cycles (Experimental): Enrolled patients may start romiplostim, as early as cycle 1 day 1; all patients MUST initiate romiplostim no later than 2 weeks from the start of the 5th cycle of chemotherapy. If plt count < 200,000/mm3, patients will start romiplostim based on their weight.
  Interventions: Drug: Romiplostim (AMG-531)

INTERVENTIONS:
Drug: Romiplostim (AMG-531) — Romiplostim may be started as supportive care, as early as cycle 1 day 1; all patients MUST initiate romiplostim no later than 2 weeks from the start of the 5th cycle of chemotherapy (see exception below for patients with platelet count of 200,000 or greater). If plt count < 200,000/mm3, patients will start romiplostim based on their weight
  Other Names: NPLATE

SUMMARY:
The goal of this clinical trial is to to assess the efficacy of romiplostim as a supportive care measure in patients with a new diagnosis of Ewing sarcoma receiving interval-compressed chemotherapy. The main questions it aims to answer are:

1. To demonstrate the efficacy of romiplostim in patients with newly diagnosed Ewing sarcoma, measured specifically as the rate of chemotherapy-induced thrombocytopenia (CIT), defined as a failure to achieve platelet recovery.
2. To determine the safety of incorporation of romiplostim supportive care when given concurrently with Ewing sarcoma therapy.
3. To determine the feasibility of incorporation of romiplostim supportive care into upfront Ewing sarcoma regimens

DETAILED DESCRIPTION:
This is a single-arm, multi-center clinical trial to assess the efficacy of romiplostim as a supportive care measure in patients with a new diagnosis of Ewing sarcoma receiving interval-compressed chemotherapy. Patients will be enrolled and started on romiplostim as early as cycle 1 day 1 of their chemotherapy, but no later than 2 weeks from the start of the 5th cycle. If their platelet count is < 200,000/mm3, patients will start romiplostim based on their weight. Dose escalation of romiplostim may occur weekly if platelet count is < 200,000/mm3. Once maximum dose of romiplostim is reached, this dose level will be maintained every 7 days (+/- 2 days).

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be >1 year old at the time of study consent.
* Diagnosis: Patients with a new diagnosis of Ewing sarcoma treated with interval-compressed chemotherapy as per AEWS0031, AEWS1221, or AEWS1031.
* Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Marrow disease: Patients with metastatic Ewing sarcoma to the bone marrow are not eligible. Marrow staging is not required for this study but should be performed if clinically indicated.
* Concomitant therapy, cancer directed: Patients receiving whole lung radiation, >50% of pelvic irradiation, other substantial bone marrow radiation (i.e. ≥ 50% of vertebral marrow space), or patients undergoing pneumonectomy as a component of local control before cycle 14, are not eligible. These therapies are not an exclusion if instituted during or after cycle 14.
* Concomitant therapy, non-cancer directed:

  * Patients requiring hematopoietic stem cell rescue are not eligible.
  * Previous use of romiplostim, eltrombopag or any other platelet-producing agent is not allowed.
  * Previous therapy for immune thrombocytopenia and related conditions, including rituximab, mycophenolic acid, protracted systemic steroids, and/or IVIG, is prohibited.
  * Treatment with erythropoietin-stimulating agents is prohibited.
  * Patients receiving another investigational drug are not eligible.
  * Patients who are receiving prophylactic dosing of heparin (i.e. enoxaparin) or oral anticoagulants (i.e. rivaroxaban) for thrombosis prevention may be considered for enrollment but will be excluded from secondary aim 'a' analysis (efficacy measured as the median platelet count and transfusion dependency) given shift in transfusion thresholds.
* Concurrent Illnesses: Patients with a history of or current diagnosis of bone marrow failure, hematologic malignancy, pro-thrombotic condition, or platelet disorder (including immune or heparin induced thrombocytopenia) are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the study (including safety monitoring requirements of the study) are not eligible.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of evaluable participants (11 or fewer of 26) that develop CIT during the continuation phase of compressed-interval chemotherapy compared to institutional historical control rate. | 52 weeks
  CIT is defined as failure to achieve platelet recovery ((≥ 75,000/µL post nadir, without transfusion, or a platelet count sufficient to resume chemotherapy per provider and institutional standard) within 7 days of planned chemotherapy cycle start, measured during the continuation phase (beyond cycle 6)
Measure adverse events with the addition of romiplostim when given with chemotherapy. | 52 weeks
  To determine the safety of incorporation of romiplostim supportive care when given concurrently with Ewing sarcoma therapy.
Number of patients able to receive the majority of planned romiplostim doses. | 52 weeks
  Feasibility will be met if fewer than 9 of 26 enrolled patients fail to receive at least 60% of planned romiplostim doses (excluding doses held for thrombocytosis or post-operatively) from initiation through at least the end of the 13th cycle of chemotherapy or through at least the end of the 16th cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Turpin, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Phoenix Children's, Phoenix, Arizona
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Womer RB, West DC, Krailo MD, Dickman PS, Pawel BR, Grier HE, Marcus K, Sailer S, Healey JH, Dormans JP, Weiss AR. Randomized controlled trial of interval-compressed chemotherapy for the treatment of localized Ewing sarcoma: a report from the Children's Oncology Group. J Clin Oncol. 2012 Nov 20;30(33):4148-54. doi: 10.1200/JCO.2011.41.5703. Epub 2012 Oct 22. PMID 23091096
- [Background] Vadhan-Raj S. Management of chemotherapy-induced thrombocytopenia: current status of thrombopoietic agents. Semin Hematol. 2009 Jan;46(1 Suppl 2):S26-32. doi: 10.1053/j.seminhematol.2008.12.007. PMID 19245931
- [Background] Tamamyan G, Danielyan S, Lambert MP. Chemotherapy induced thrombocytopenia in pediatric oncology. Crit Rev Oncol Hematol. 2016 Mar;99:299-307. doi: 10.1016/j.critrevonc.2016.01.005. Epub 2016 Jan 15. PMID 26811139
- [Background] Womer RB, Daller RT, Fenton JG, Miser JS. Granulocyte colony stimulating factor permits dose intensification by interval compression in the treatment of Ewing's sarcomas and soft tissue sarcomas in children. Eur J Cancer. 2000 Jan;36(1):87-94. doi: 10.1016/s0959-8049(99)00236-1. PMID 10741300
- [Background] Weycker D, Hatfield M, Grossman A, Hanau A, Lonshteyn A, Sharma A, Chandler D. Risk and consequences of chemotherapy-induced thrombocytopenia in US clinical practice. BMC Cancer. 2019 Feb 14;19(1):151. doi: 10.1186/s12885-019-5354-5. PMID 30764783
- [Background] Bracho F, Krailo MD, Shen V, Bergeron S, Davenport V, Liu-Mares W, Blazar BR, Panoskaltsis-Mortari A, van de Ven C, Secola R, Ames MM, Reid JM, Reaman GH, Cairo MS. A phase I clinical, pharmacological, and biological trial of interleukin 6 plus granulocyte-colony stimulating factor after ifosfamide, carboplatin, and etoposide in children with recurrent/refractory solid tumors: enhanced hematological responses but a high incidence of grade III/IV constitutional toxicities. Clin Cancer Res. 2001 Jan;7(1):58-67. PMID 11205919
- [Background] Cairo MS, Davenport V, Bessmertny O, Goldman SC, Berg SL, Kreissman SG, Laver J, Shen V, Secola R, van de Ven C, Reaman GH. Phase I/II dose escalation study of recombinant human interleukin-11 following ifosfamide, carboplatin and etoposide in children, adolescents and young adults with solid tumours or lymphoma: a clinical, haematological and biological study. Br J Haematol. 2005 Jan;128(1):49-58. doi: 10.1111/j.1365-2141.2004.05281.x. PMID 15606549
- [Background] Angiolillo AL, Davenport V, Bonilla MA, van de Ven C, Ayello J, Militano O, Miller LL, Krailo M, Reaman G, Cairo MS; Children's Oncology Group. A phase I clinical, pharmacologic, and biologic study of thrombopoietin and granulocyte colony-stimulating factor in children receiving ifosfamide, carboplatin, and etoposide chemotherapy for recurrent or refractory solid tumors: a Children's Oncology Group experience. Clin Cancer Res. 2005 Apr 1;11(7):2644-50. doi: 10.1158/1078-0432.CCR-04-1959. PMID 15814645
- [Background] Li J, Yang C, Xia Y, Bertino A, Glaspy J, Roberts M, Kuter DJ. Thrombocytopenia caused by the development of antibodies to thrombopoietin. Blood. 2001 Dec 1;98(12):3241-8. doi: 10.1182/blood.v98.12.3241. PMID 11719360
- [Background] Kuter DJ. Milestones in understanding platelet production: a historical overview. Br J Haematol. 2014 Apr;165(2):248-58. doi: 10.1111/bjh.12781. Epub 2014 Feb 14. PMID 24528208
- [Background] Zhang J, Liang Y, Ai Y, Xie J, Li Y, Zheng W. Thrombopoietin-receptor agonists for children with immune thrombocytopenia: a systematic review. Expert Opin Pharmacother. 2017 Oct;18(15):1543-1551. doi: 10.1080/14656566.2017.1373091. Epub 2017 Sep 4. PMID 28845713
- [Background] Tumaini Massaro J, Chen Y, Ke Z. Efficacy and safety of thrombopoietin receptor agonists in children with chronic immune thrombocytopenic purpura: meta-analysis. Platelets. 2019;30(7):828-835. doi: 10.1080/09537104.2019.1572873. Epub 2019 Feb 27. PMID 30810479
- [Background] Bowers C, Mytych DT, Lawrence T, Wang K, Barger TE, Eisen M, Bennett CM, Tarantino MD. Assessment of romiplostim immunogenicity in pediatric patients in clinical trials and in a global postmarketing registry. Blood Adv. 2021 Dec 14;5(23):4969-4979. doi: 10.1182/bloodadvances.2021005105. PMID 34638135
- [Background] Mones JV, Soff G. Management of Thrombocytopenia in Cancer Patients. Cancer Treat Res. 2019;179:139-150. doi: 10.1007/978-3-030-20315-3_9. PMID 31317485
- [Background] Al-Samkari H, Soff GA. Clinical challenges and promising therapies for chemotherapy-induced thrombocytopenia. Expert Rev Hematol. 2021 May;14(5):437-448. doi: 10.1080/17474086.2021.1924053. Epub 2021 May 13. PMID 33926362
- [Background] Jacobson AE, Shah N, Setty BA. Romiplostim for therapy-related thrombocytopenia in pediatric malignancies. Pediatr Blood Cancer. 2017 Aug;64(8). doi: 10.1002/pbc.26473. Epub 2017 Feb 2. PMID 28150377
- [Background] Merjaneh N, Young J, Mangoli A, Olsen M, Setty B, Lane A, Nagarajan R, Pressey JG, Turpin B. Chemotherapy-induced thrombocytopenia in Ewing sarcoma: Implications and potential for romiplostim supportive care. Pediatr Blood Cancer. 2022 Jul;69(7):e29548. doi: 10.1002/pbc.29548. Epub 2021 Dec 28. PMID 34962714
- [Background] Tarantino MD, Bussel JB, Blanchette VS, Despotovic J, Bennett C, Raj A, Williams B, Beam D, Morales J, Rose MJ, Carpenter N, Nie K, Eisen M. Romiplostim in children with immune thrombocytopenia: a phase 3, randomised, double-blind, placebo-controlled study. Lancet. 2016 Jul 2;388(10039):45-54. doi: 10.1016/S0140-6736(16)00279-8. Epub 2016 Apr 18. PMID 27103127
- [Background] Al-Samkari H, Kuter DJ. Thrombopoietin level predicts response to treatment with eltrombopag and romiplostim in immune thrombocytopenia. Am J Hematol. 2018 Dec;93(12):1501-1508. doi: 10.1002/ajh.25275. Epub 2018 Sep 26. PMID 30187942
- [Background] Song AB, Goodarzi K, Karp Leaf R, Kuter DJ, Al-Samkari H. Thrombopoietin level predicts response to treatment with romiplostim in chemotherapy-induced thrombocytopenia. Am J Hematol. 2021 Dec 1;96(12):1563-1568. doi: 10.1002/ajh.26338. Epub 2021 Sep 10. PMID 34453757
- [Background] Xie Z, Zeidan AM. CHIPing away the progression potential of CHIP: A new reality in the making. Blood Rev. 2023 Mar;58:101001. doi: 10.1016/j.blre.2022.101001. Epub 2022 Aug 15. PMID 35989137
- [Background] Giagounidis A, Mufti GJ, Fenaux P, Sekeres MA, Szer J, Platzbecker U, Kuendgen A, Gaidano G, Wiktor-Jedrzejczak W, Hu K, Woodard P, Yang AS, Kantarjian HM. Results of a randomized, double-blind study of romiplostim versus placebo in patients with low/intermediate-1-risk myelodysplastic syndrome and thrombocytopenia. Cancer. 2014 Jun 15;120(12):1838-46. doi: 10.1002/cncr.28663. Epub 2014 Apr 4. PMID 24706489
- [Background] Vishnu P, Aboulafia DM. Long-term safety and efficacy of romiplostim for treatment of immune thrombocytopenia. J Blood Med. 2016 May 25;7:99-106. doi: 10.2147/JBM.S80646. eCollection 2016. PMID 27307776
- [Background] Wilkins CR, Ortiz J, Gilbert LJ, Yin S, Mones JV, Parameswaran R, Mantha S, Soff GA. Romiplostim for chemotherapy-induced thrombocytopenia: Efficacy and safety of extended use. Res Pract Thromb Haemost. 2022 May 10;6(3):e12701. doi: 10.1002/rth2.12701. eCollection 2022 Mar. PMID 35582038
- [Background] Soff GA, Miao Y, Bendheim G, Batista J, Mones JV, Parameswaran R, Wilkins CR, Devlin SM, Abou-Alfa GK, Cercek A, Kemeny NE, Sarasohn DM, Mantha S. Romiplostim Treatment of Chemotherapy-Induced Thrombocytopenia. J Clin Oncol. 2019 Nov 1;37(31):2892-2898. doi: 10.1200/JCO.18.01931. Epub 2019 Sep 23. PMID 31545663
- [Background] Al-Samkari H, Parnes AD, Goodarzi K, Weitzman JI, Connors JM, Kuter DJ. A multicenter study of romiplostim for chemotherapy-induced thrombocytopenia in solid tumors and hematologic malignancies. Haematologica. 2021 Apr 1;106(4):1148-1157. doi: 10.3324/haematol.2020.251900. PMID 32499239
- [Background] Paz-Priel I, Long L, Helman LJ, Mackall CL, Wayne AS. Thromboembolic events in children and young adults with pediatric sarcoma. J Clin Oncol. 2007 Apr 20;25(12):1519-24. doi: 10.1200/JCO.2006.06.9930. PMID 17442994
- [Background] Athale U, Cox S, Siciliano S, Chan AK. Thromboembolism in children with sarcoma. Pediatr Blood Cancer. 2007 Aug;49(2):171-6. doi: 10.1002/pbc.21047. PMID 16991135